CLINICAL TRIAL: NCT05201963
Title: Effect of Ultrasound Guided Erector Spinae Plane Block Versus Ultrasound Guided Serratus Anterior Block on the Incidence of Post Mastectomy Pain Syndrome, Randomized Double Blinded Controlled Study
Brief Title: Erector Spinae Plane Block Versus Serratus Anterior Block on Post Mastectomy Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Mohammed Magdy Abdelrahman Elsayed, Assistant Lecturer of Anesthesiology , ICU and Pain Management, National Cancer Institute, Egypt
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AP2110-30111
Record Dates: First submitted 2021-12-22; First posted 2022-01-21 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer; Post-mastectomy Pain Syndrome; Acute Pain
Keywords: Breast Cancer; Post Mastectomy Pain Syndrome; Erector Spinae Plane Block; Serratus Anterior Plane Block
MeSH Terms: conditions — Breast Neoplasms; Acute Pain

STUDY DESIGN:
Intervention Model Description: The patients will be randomly assigned into 3 equal groups using computer generated random numbers in opaque closed envelopes, each of which will include 40 patients. Group 1 control group N=40, Group 2 ((Serratus Anterior Plane Block SAPB)) N=40 Patients will receive Ultrasound guided Serratus Anterior Plane Block with injection of 30 ml levobupivacaine 0.25% and Group 3 ((Erector Spinae Plane Block ESB)) N=40 Patients will receive Ultrasound guided erector spinae plane block with injection of 30 ml levobupivacaine 0.25%. Randomization will be done by a statistician and each group of the patient will be revealed only when the included patient is transferred to the preanesthetic room.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 control group (No Intervention): Control group will recive only IV Opioids
- Group 2 ((Serratus Anterior Plane Block SAPB)) (Experimental): Patients will receive Ultrasound guided Serratus Anterior Plane Block with injection of 30 ml levobupivacaine 0.25%
  Interventions: Procedure: Serratus Anterior Plane Block
- Group 3 ((Erector Spinae Plane Block ESB)) (Experimental): Patients will receive Ultrasound guided erector spinae plane block with injection of 30 ml levobupivacaine 0.25%.
  Interventions: Procedure: Erector Spinae Plane Block

INTERVENTIONS:
Procedure: Serratus Anterior Plane Block — Full aseptic precautions applied. Ultrasound probe will be placed on the patient's midaxillary line in the longitudinal plane (lateral position with arm abduction), at the level of 5th rib, the indicator oriented toward the operator's left. With the rib, pleural line, overlying serratus anterior and latissimus dorsi muscles visualized, then, a 38-mm 22-gauge regional block needle will be advanced in-plane at an angle of approximately 45 degrees towards the 5th rib. After aspiration to avoid intravascular injection 30ml of levobupivacaine 0.25% will be injected anteriorly to the rib and deep to the serratus anterior muscle. The entirety of the needle should be visualized at all times throughout the procedure.6-13-MHz, linear transducer set for small parts and a depth of 1-4 cm is used for this block(15-16).
  Arms: Group 2 ((Serratus Anterior Plane Block SAPB))
Procedure: Erector Spinae Plane Block — Full aseptic precautions applied. Ultrasound probe will be placed on the back in a transverse orientation to identify the tip of the T5 transverse process. The tip of the transverse process will be centered on the ultrasound screen and the probe will then be rotated into a longitudinal orientation to produce a parasagittal view, in which skin, subcutaneous tissue, trapezius and erector spinae muscle will be visible superficial to T5 transverse process. Echogenic block needle will be inserted in- plane to the ultrasound beam in a cranial-to-caudal direction until contact is made with the T5 transverse process. Correct location of the needle tip in the fascial plane deep to erector spinae muscle will be confirmed by injecting 0.5-1 ml normal saline . After aspiration to avoid intravascular injection 30 ml levobupivacaine 0.25% will be performed. 6-13-MHz, linear transducer set for small parts and a depth of 4-6 cm will be used
  Arms: Group 3 ((Erector Spinae Plane Block ESB))

SUMMARY:
Breast cancer is the most common malignancy among females. Nearly 40-60% of breast surgery patients experience severe acute postoperative pain, with severe pain persisting for 6-12 months in almost 20-50% of patients (post mastectomy pain syndrome) which is defined according to International Association for the Study of Pain (IASP) as pain which persists more than 3 months after mastectomy/lumpectomy affecting the anterior thorax, axilla, and/or medial upper arm. Regionale anesthesia is one of the strategies with the potential to prevent the development of chronic pain following breast surgery. We hypothesize that erector spinae plane block is going to be more effective than serratus anterior plane block in the prevention of postmastectomy pain syndrome.

DETAILED DESCRIPTION:
Background and Rationale:

Breast cancer is the most common malignancy among females with incidence of about 2.1 million women each year. It is the most common cause for cancer-related deaths among women. (1) Modified Radical Mastectomy (MRM) is one of the main surgical treatments of breast cancer. It is account for 31% of all breast surgery cases (2). Nearly 40-60% of breast surgery patients experience severe acute postoperative pain, with severe pain persisting for 6-12 months in almost 20-50% of patients (post mastectomy pain syndrome)(3-4). Pain can be severe enough to cause long-term disabilities and interfere with sleep and performance of daily activities leading to complications such as: shoulder adhesive capsulitis (frozen shoulder), complex regional pain syndrome (causalgia) and altered sensation creating an economic burden for the health care system (5-8).

The International Association for the Study of Pain (IASP) defines PMPS as pain which persists more than 3 months after mastectomy/lumpectomy affecting the anterior thorax, axilla, and/or medial upper arm.It usually describes as feeling of burning, stabbing, and pulling around the treatment side(9) The underlying pathophysiology of PMPS is highly complicated and entangle both peripheral and central sensitization. Multiple risk factors involved in the development of PMPS including Acute postoperative pain ,Age < 40 years , Increased BMI ,Diagnosis at later-stage disease , Psychosocial factors (i.e., anxiety, depression, sleep disturbances, catastrophizing) Preoperative pain and Adjuvant therapy (chemotherapy, radiation therapy(10). Like other neuropathic pain conditions, the treatment is a difficult task (11), so the focus of current research is on perioperative measures that can mitigate the modifiable risk factors for PMPS and thereby prevent patients from developing PMPS in the first place. Recognizing the importance of postoperative pain management, a number of studies have looked at strategies with the potential to prevent the development of chronic pain following breast surgery including regional anesthesia. (12)

These regional techniques include: Intercostal nerve block, Pectoral nerve Blocks (PECI & PECS II) , Serratus Anterior Plane block (SAPB) and Erector Spinae Plane Block (ESPB). (14) Hypothesis: We hypothesize that Ultrasound guided erector spinae plane block is going to be more effective than ultrasound guided serratus anterior plane block in the prevention of postmastectomy pain syndrome in patients undergoing MRM as the injected local anesthetics acts on the dorsal and ventral rami of the thoracic spinal nerves and, thus, it is expected to block the sympathetic fibers leading to effective management of somatic and visceral pain.

Objectives:

The aim of this study is to evaluate the impact of US guided ESPB compared to US guided SAPB on the emergence of PMPS in patients undergoing MRM for cancer breast.

Study Design :

Randomized Double Blinded Controlled Study.

Population of study: 120 Female patients ASA II ,III scheduled for modified radical mastectomy under general anesthesia.

Study location: National Cancer Institute Cairo University after approval by the institutional review board.

Randomization: The patients will be randomly assigned into 3 equal comparable groups using computer generated random numbers in opaque closed envelopes, each of which will include 40 patients. Group 1 control group N=40, Group 2 ((Serratus Anterior Plane Block SAPB)) N=40.Randomization will be done by a statistician and each group of the patient will be revealed only when the included patient is transferred to the preanesthetic room.

Study Protocol: Patient assessment; History, physical exam, laboratory and radiological investigations at preoperative assessment clinic National Cancer Institute Cairo University. Preoperative assessment at night of surgery. The patients will be instructed how to report pain by means of Numeric Pain Rating Scale, in which 0 = no pain and 10 =worst possible pain. Informed consent will be obtained, base line Flanagan Quality of Life Scale (QOLS) and Barthel Activities of Daily Living scale (ADL) will be obtained.Preoperative fasting; minimum of 6 hours for food and minimum of 2 hours for water and clear fluids.20G IV cannula will be inserted. All patients will be premedicated with IV midazolam 0.01-0.02 mg\kg 30 minutes preoperatively.

Anesthetic Management:

Monitoring: all patients will be monitored continuously using ECG, NIBP, peripheral arterial oxygen saturation and end tidal carbon dioxide throughout the duration of surgery. Regimen of IV 2 μg/kg fentanyl and propofol IV 2 mg /kg will be used for Induction of general anaesthesia. Tracheal intubation will be facilitated using 0.5 mg/kg IV of rocuronium.

After Induction of GA group 2 patients will receive serratus anterior plane block and patients of group 3 will receive erector spinae plane block. Both blocks will be done with the patients at lateral position.

In both blocks Fujifilm Sonosite M-Turbo Ultrasound system will be used.

After performing blocks lung ultrasound is performed to exclude pneumothorax, chest is divided to 6 quadrants: Anterior upper and anterior lower quadrants Lateral upper and lower quadrants Posterior upper and lower quadrants All quadrants will be scanned especially upper quadrants looking for signs of pneumothorax such as absence of lung sliding, presence of B lines, barcode or stratosphere sign and lungpoint sign. Lung ultrasound will be done after performing block and post operative at PACU (18).

Anaesthesia will be maintained with inhaled sevoflurane 2-2.5% in oxygen enriched air (FiO2=0.5). Maintenance doses of rocuronium o.1 m\kg will be provided every 30 minutes. Paracetamol 1000 mg and IV ketorolac 30mg will be provided as a part of multimodal analgesia. Rescue analgesia of fentanyl 1 μg/kg will be given if the mean arterial blood pressure or heart rate rises above 20% of baseline levels. Ringer acetate will be infused to replace their fluid deficit, maintenance and losses, and the patients will be mechanically ventilated at appropriate settings that keep end-tidal CO2 at 30- 35 mmHg. 1st reading of mean arterial pressure (MAP) and heart rate (HR) will be recorded before induction of general anaesthesia to be defined as a baseline reading another reading will be noted immediately before surgical incision and at 30-minute intervals intraoperatively. At the end of surgery residual neuromuscular blockade will be reversed using neostigmine (0.05 mg/kg) and atropine (0.02 mg/kg), and extubation will be performed after complete recovery of the airway reflexes. The patients will be transferred to the post-anaesthesia care unit (PACU) where the, Numeric Pain Rating Scale score, MAP and heart rate will be noted immediately on arrival, where they will be observed for 2 hours then discharged to the ward. Lung ultrasound will be performed once again at PACU looking for signs of pneumothorax. Rescue analgesia will be provided in the form of IV morphine 3 mg boluses if the patient indicates Numeric Pain Rating Scale ≥ 4. The total amount of morphine given in 24 hours will be recorded for the 3 groups. A maximum dose of 0.5 mg/kg/24hours of morphine is allowed. Thereafter, the patients will be shifted to their respective ward, Multimodal analgesia will be provided as the following: IV paracetamol 1000mg \8 hours IV ketorolac 30mg\8 hours. There, Numeric Pain Rating Scale score, MAP and heart rate will be noted at 4, 8, 12, 16, 20 and 24 hours postoperatively. Side effects such as nausea, vomiting, sedation and respiratory depression (respiratory rate <10/minute) will be recorded. Postoperative nausea and vomiting (PONV) will be rated on a four-point verbal scale and 0.1 mg/kg of IV ondansetron will be given to patients with moderate or severe postoperative nausea and vomiting. (19) Sedation will be assessed with Ramsay score(20).

On discharge from the hospital, analgesia is going to be provided in the form of oral/parenteral paracetamol, NSAIDs and tramadol HCl according to patient preference and drugs availability for the rest of the 1st postoperative week. Average daily drug consumption after discharge will be recorded. Patients will be evaluated at the follow-up by phone call or interview at the pain clinic on 2,4,8,12 and 24 postoperative weeks. NPRS will be recorded daily in the 1st week and then at 2, 4, 8 ,12 and 24 weeks postoperttively. Neuropathic pain will be evaluated according to the Grading System for Neuropathic Pain (GSNP). Positive neuropathic cases are those with GSNP 3 (probable) or GSNP 4 (definite) i.e. GSNP ≥ 3 .(21). Flanagan Quality of Life Scale (QOLS) will be used for Quality of life assessemnt, The scale will be explained to the patients and the total score will calculated and recorded at the preoperative assessment (baseline) and at postoperative weeks 2, 3, 4, 8 ,12 and 24(22).Barthel Activities of Daily Living scale (ADL) is going to be used to record patients activity level at postoperative weeks 2, 3, 4, 8 ,12 and 24 (23).

PMPS is defined as neuropathic pain which persists more than 3 months after mastectomy/lumpectomy affecting the anterior thorax, axilla, and/or medial upper arm(9).

Patients who are going to develop post-mastectomy neuropathic pain will treated by the following regimen according to local protocol at the NCI CU: pregabalin 75-300 mg/day and amitriptyline 10-25 mg/day. Analgesics such as paracetamol, NSAIDs, tramadol HCl 100-400 mg/day and oxycodone 20-60 mg/day will be added if required according to pain severity.

Sample Size:

As there is no study addressed the same research question in these cases. Sample size was calculated according to a preliminary analysis of the first 63 patients (21 in each group) as a pilot to detect the proportion of PMPS in each group, 61% of group 1 patients developed PMPS compared to 42% and 28% in group 2 and 3 respectively. To achieve 95% confidence level a minimum sample size of 33 patients per group will be needed. To compensate for possible losses 15% will be added, 120 Patients in total will be recruited (40 per group).

Statistical analysis:

SPSS version 27.0 will be used in data analysis. Quantitative variables will be tested for normality to select appropriate statistical tests. Quantitative variables will be described as mean +- standard deviation or median and range.Comparison of of two independent groups will be done using t test or non parametric Mann Whittney u test . Data including more two groups will be tested using either by ANOVA or non parametric Kruskal-Wallis test.Post-hoc test will be used for pairwise comparisons and will be Tucky adjusted. Chi-square and Fisher Exact are going to be used for testing qualitative data . P is going to be always two tailed and set significant at 0.05 level.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* Type of surgery; Modified Radical Mastectomy MRM
* Physical status ASA II, III.
* Body mass index (BMI): > 20 kg/m2 and < 35 kg/m2.

Exclusion Criteria:

* Patient refusal.
* BMI <20 kg/m2 and >35 kg/m2
* Known sensitivity or contraindication to drug used in the study (local anaesthetics, opioids).
* History of psychological disorders and/or chronic pain.
* Contraindication to regional anaesthesia e.g. local sepsis, pre- existing peripheral neuropathies and coagulopathy.
* Severe respiratory or cardiac disorders. Advanced liver or kidney disease.
* Pregnancy.
* Physical status ASA IV and Male patients.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Incidence of patients developing PMPS. | 6 months
  Number and Percentage of patients developing PMPS

SECONDARY OUTCOMES:
Patient's Quality of life according to Flanagan Quality of Life Scale (QOLS) | 6 motnths
  Flanagan Quality of Life Scale (QOLS) will be used for Quality of life assessemnt, which is a 16-item (domain) questionnaire with each item scored from 1 to 7 points. The scale will be explained to the patients and the total score will calculated and recorded at the preoperative assessment (baseline) and at postoperative weeks 2, 3, 4, 8 ,12 and 24
Severity of PMPS according to Grading system for neuropathic pain (GSNP) | 6 motnths
  Neuropathic pain will be evaluated according to the Grading System for Neuropathic Pain (GSNP). Positive neuropathic cases are those with GSNP 3 (probable) or GSNP 4 (definite) i.e. GSNP ≥ 3 . Grading system for neuropathic pain (GSNP) is as follows: Grade 1 (unlikely), Grade 2 (possible), Grade 3 (probable), and Grade 4 (definite )
Postoperative Patient's activity level according to Barthel Activities of Daily Living Scale ADL | 6 months
  Barthel Activities of Daily Living scale (ADL) is going to be used to record patients activity level at postoperative weeks 2, 3, 4, 8 ,12 and 24. This scale comprises 10 basic daily activities (bowel, bladder, feeding, toilet, bathing, dressing, grooming, walking, stairs and transfer) with each item scored as 0 = need complete help, 1 = need some help or 2 = need no help
Total amount of morphine consumed postoperatively | 24 hours
  Total amount of morphine consumed postoperatively in mg
Total amount of fentanyl consumed intraoperative | Time of surgry
  Total amount of fentanyl consumed intraoperative in mcg
Change in heart rate intraoperative | 24 hours
  Change in heart rate intraoperative in beat\min
Change in Mean Artertial Blood Pressure (MAP) intraoperative | 24 hours
  Change in Mean Artertial Blood Pressure (MAP) intraoperative in mmHg
The degree of postoperative sedation according to Ramsay scores. | 24 hours
  Sedation will be assessed with Ramsay score (1 = anxious or restless or both; 2 = cooperative, orientated, and tranquil; 3= responding to commands; 4 = brisk response to stimulus; 5 = sluggish response to stimulus; and 6 = no response to stimulus). A Ramsay score of 5 or 6 will be considered excessively high sedation levels; a Ramsay score of 2 to 4 will be considered adequate sedation levels needing observation; a Ramsay score of 1 will be considered inadequate or insufficient sedation Levels
Postoperative nausea and vomiting (PONV). | 24 hours
  Postoperative nausea and vomiting (PONV) will be rated on a four-point verbal scale; (none =no nausea, mild =nausea but no vomiting, moderate=vomiting one attack, severe =vomiting >one attack). 0.1 mg/kg of IV ondansetron will be given to patients with moderate or severe postoperative nausea and vomiting.
Change in heart rate postoperatively. | 24 hours
  Change in heart rate postoperatively in beat\min.
Change in Mean Artertial Blood Pressure (MAP) postoperatively. | 24 hours
  Change in Mean Artertial Blood Pressure (MAP) postoperatively in mmHg.
Time of first rescue analgesia. | 24 hours
  1st time the patient asks for analgesia or 1st time when NPRS equal to or more than 10
Complications related to blocks | 24 hours
  Number of patinets developing complications related to blocks such as local anaesthetic systemic toxicity, pneumothorax and arterial puncture.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Magdy, Master, Principal Investigator — National Cancer Institute Cairo University; Somaya Elsheikh Abdelaziz, Professor, Study Chair — National Cancer Institute Cairo University; Ahmed H. Bekir, Professor, Study Director — National Cancer Institute Cairo University; Sayed M. Abed, Lecturer, Study Director — National Cancer Institute Cairo University; Mohammed ElSaed Abdelfattah, Lecturer, Study Director — National Cancer Institute Cairo University
Locations (1):
- National Cancer Institute, Cairo, Cairo Governorate, Egypt

REFERENCES:
- [Background] Garg R, Bhan S, Vig S. Newer regional analgesia interventions (fascial plane blocks) for breast surgeries: Review of literature. Indian J Anaesth. 2018 Apr;62(4):254-262. doi: 10.4103/ija.IJA_46_18. PMID 29720750
- [Background] De Cassai A, Bonvicini D, Correale C, Sandei L, Tulgar S, Tonetti T. Erector spinae plane block: a systematic qualitative review. Minerva Anestesiol. 2019 Mar;85(3):308-319. doi: 10.23736/S0375-9393.18.13341-4. Epub 2019 Jan 4. PMID 30621377
- [Background] Gong Y, Tan Q, Qin Q, Wei C. Prevalence of postmastectomy pain syndrome and associated risk factors: A large single-institution cohort study. Medicine (Baltimore). 2020 May;99(20):e19834. doi: 10.1097/MD.0000000000019834. PMID 32443289
- [Background] Smith WC, Bourne D, Squair J, Phillips DO, Chambers WA. A retrospective cohort study of post mastectomy pain syndrome. Pain. 1999 Oct;83(1):91-5. doi: 10.1016/s0304-3959(99)00076-7. PMID 10506676
- [Background] Miguel R, Kuhn AM, Shons AR, Dyches P, Ebert MD, Peltz ES, Nguyen K, Cox CE. The effect of sentinel node selective axillary lymphadenectomy on the incidence of postmastectomy pain syndrome. Cancer Control. 2001 Sep-Oct;8(5):427-30. doi: 10.1177/107327480100800506. PMID 11579339
- [Background] Caffo O, Amichetti M, Ferro A, Lucenti A, Valduga F, Galligioni E. Pain and quality of life after surgery for breast cancer. Breast Cancer Res Treat. 2003 Jul;80(1):39-48. doi: 10.1023/A:1024435101619. PMID 12889597
- [Background] Fecho K, Miller NR, Merritt SA, Klauber-Demore N, Hultman CS, Blau WS. Acute and persistent postoperative pain after breast surgery. Pain Med. 2009 May-Jun;10(4):708-15. doi: 10.1111/j.1526-4637.2009.00611.x. Epub 2009 Apr 22. PMID 19453965
- [Background] Capuco A, Urits I, Orhurhu V, Chun R, Shukla B, Burke M, Kaye RJ, Garcia AJ, Kaye AD, Viswanath O. A Comprehensive Review of the Diagnosis, Treatment, and Management of Postmastectomy Pain Syndrome. Curr Pain Headache Rep. 2020 Jun 11;24(8):41. doi: 10.1007/s11916-020-00876-6. PMID 32529416
- [Background] Larsson IM, Ahm Sorensen J, Bille C. The Post-mastectomy Pain Syndrome-A Systematic Review of the Treatment Modalities. Breast J. 2017 May;23(3):338-343. doi: 10.1111/tbj.12739. Epub 2017 Jan 30. PMID 28133848
- [Background] Tait RC, Zoberi K, Ferguson M, Levenhagen K, Luebbert RA, Rowland K, Salsich GB, Herndon C. Persistent Post-Mastectomy Pain: Risk Factors and Current Approaches to Treatment. J Pain. 2018 Dec;19(12):1367-1383. doi: 10.1016/j.jpain.2018.06.002. Epub 2018 Jun 30. PMID 29966772
- [Background] Blanco R. The 'pecs block': a novel technique for providing analgesia after breast surgery. Anaesthesia. 2011 Sep;66(9):847-8. doi: 10.1111/j.1365-2044.2011.06838.x. No abstract available. PMID 21831090
- [Background] Blanco R, Parras T, McDonnell JG, Prats-Galino A. Serratus plane block: a novel ultrasound-guided thoracic wall nerve block. Anaesthesia. 2013 Nov;68(11):1107-13. doi: 10.1111/anae.12344. Epub 2013 Aug 7. PMID 23923989
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Lichtenstein DA. BLUE-protocol and FALLS-protocol: two applications of lung ultrasound in the critically ill. Chest. 2015 Jun;147(6):1659-1670. doi: 10.1378/chest.14-1313. PMID 26033127
- [Background] Apfel CC, Kranke P, Eberhart LH, Roos A, Roewer N. Comparison of predictive models for postoperative nausea and vomiting. Br J Anaesth. 2002 Feb;88(2):234-40. doi: 10.1093/bja/88.2.234. PMID 11883387